CLINICAL TRIAL: NCT03644173
Title: Personal Resilience Empowerment Program (PREP) in the Perioperative Setting of Surgically Treated Cancer Patients
Brief Title: Personal Resilience Empowerment Program Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB#201801121J
Record Dates: First submitted 2018-08-20; First posted 2018-08-23 (Actual); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Lung Cancer; Cholangiocarcinoma; Pancreatic Cancer; Liver Cancer
Keywords: integrative medicine; cancer patients
MeSH Terms: conditions — Lung Neoplasms; Cholangiocarcinoma; Pancreatic Neoplasms; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study arm - PREP Intervention (Experimental): Participants receiving the coaching intervention
  Interventions: Behavioral: Personal Resilience Empowerment Program including 5 sessions with health coaches

INTERVENTIONS:
Behavioral: Personal Resilience Empowerment Program including 5 sessions with health coaches — 5 coaching sessions that will take place either in-person or over the phone with a research nurse (RN)-Health Coach. During the sessions, the health coach will focus on introducing the 5 pillars of health and well-being: sleep, activity, purpose, nutrition and resilience. Will introduce breathing techniques participants and will teach patients how to acquire mind-body skills to assist in stress management, learn to thrive by building resilience, feel empowered to manage their health, gain self-care skills to decrease anxiety, pain and nausea naturally, control the stress response and trigger the relaxation response to promote well-being and discover what foods fuel the body in preparation for healing, during recovery and overall health.

SUMMARY:
The Personal Resilience Empowerment Program (PREP) at Hackensack Meridian Integrative Health & Medicine was designed in Legacy Meridian to assist all selected patients with upcoming hospitalization. For the "Personal Resilience Empowerment Program (PREP) in the perioperative setting of surgically treated cancer patients", hereafter "the Project or PREP", the Hackensack Meridian Integrative Health & Medicine is designing a new pilot program to focus on the needs of oncology patients.

All patients diagnosed with cancer that will undergo a scheduled surgical (Hepato-Biliary, and Thoracic) procedure in Hackensack Meridian Health and specifically in the Jersey Shore University Medical Center, will be eligible to participate (for more details please see eligibility criteria, section 4).

Overall, this pilot project will include 5 coaching sessions and an introductory session/visit that will take place on the physician's office. The initial physician visit will focus on patient eligibility, introduction to the Project, informed consent and a pre-intervention survey and will be conducted by the principal investigator or one of the sub-investigators listed above. The following 5 sessions will be conducted by one of the integrative health coaches/registered nurses (for details please see section 5). A post-intervention survey will be completed during the final session and repeated at one month, and at 3 months from the final session.

The goal of this project is to investigate whether using the PREP as an intervention in patients diagnosed with cancer would result in improving various metrics including improvements to resilience, sleep, activity, purpose, nutrition, empowerment to manage one's own health and well-being, decrease in pain medication use and more rapid return to previous functional status according to Eastern Cooperative Oncology Group (ECOG).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cancer of the thoracic (lung), hepatobiliary system (cholangiocarcinoma, pancreatic, liver) that will undergo a scheduled surgical procedure
* Able to understand and sign the informed consent form
* Willingness to participate in the study and comply with protocol requirements

Exclusion Criteria:

* Unable to provide consent
* Unable to participate at the discretion of the PI based on the ECOG survey (if ECOG >1). See section 5 and appendix 1 for details.
* Non- English speaking patients .
* Opioid use for non-malignant pain for greater than 7 days 6 Terminal or Stage 4 cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Matteotti, MD, Principal Investigator — Hackensack Meridian Health
Locations (2):
- United States (2):
  - Hackensack Meridian Health - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Hackensack Meridian Health - Riverview Medical Center, Red Bank, New Jersey

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Personal Resilience Empowerment Program: Participants who were enrolled and completed all visits
Period: Participants at Last Visit (Pre-surveys)
Arm/Group | Personal Resilience Empowerment Program
Started | 37
Completed | 16
Not Completed | 21
Not completed — Lost to Follow-up | 21
Period: Participants at the 1-month Follow up
Arm/Group | Personal Resilience Empowerment Program
Started | 16
Completed | 12
Not Completed | 4
Not completed — Lost to Follow-up | 2
Not completed — Death | 2
Period: Participants at the 3-month Follow up
Arm/Group | Personal Resilience Empowerment Program
Started | 12
Completed | 10
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Participants who completed the visits (even if they did not complete the follow-up surveys)
Groups:
- Personal Resilience Empowerment Program: Participants who were enrolled and attended at least one visit
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 10
Age, Continuous [Mean (Full Range); unit: years] | 67.68 [38 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Sleep
Description: Quality of life concerning sleep (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the post intervention survey
Time Frame: Within two weeks from discharge, following the the post-operative visit (during the same day they would have the post-op visit, last coaching session and the post-intervention survey)
Population: Change in the question regarding sleep (t-test) between the pre and the post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 16
scores on a scale
  7-8 hours of sleep/day | -1.06 (1.95)
  Waking up rested: number analyzed (Participants) | 15
  Waking up rested | -0.80 (1.97)

2. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Activity
Description: Quality of life concerning activity (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the post intervention survey
Time Frame: as for outcome 1
Population: Change in the question regarding activity (t-test) between the pre and the post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 16
scores on a scale
  Remaining physically active | -0.13 (1.78)
  Needing help with everyday activities | 0.56 (1.90)

3. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Purpose
Description: Quality of life concerning feeling of purpose (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the post intervention survey
Time Frame: as for outcome 1
Population: Change in the question regarding activity (t-test) between the pre and the post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 16
scores on a scale | -0.19 (0.66)

4. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Nutrition
Description: Quality of life concerning nutrition (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the post intervention survey
Time Frame: as for outcome 1
Population: Change in the question regarding activity (t-test) between the pre and the post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 15
scores on a scale
  5-10 servings of fruits/day | 0.60 (1.40)
  Avoiding fast food | 1.00 (1.56)

5. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Sleep
Description: Quality of life concerning sleep (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre-intervention survey and 1-month post intervention survey
Time Frame: At 1 month Post intervention (survey was sent at 30 days after the last couching session)
Population: Change in the question regarding sleep (t-test) between the pre and the 1-month post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 12
scores on a scale
  7-8 hours of sleep/day | -0.33 (1.23)
  Waking up rested | 0.08 (1.16)

6. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Activity
Description: Quality of life concerning activity (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the 1-month post intervention survey
Time Frame: At 1 month Post intervention (survey was sent at 30 days after the last couching session)
Population: Change in the question regarding activity (t-test) between the pre and the post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 12
scores on a scale
  Remaining physically active | 0.67 (1.23)
  Needing help with everyday activities | -0.08 (1.73)

7. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Purpose
Description: Quality of life concerning feeling of purpose (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the 1-month post intervention survey
Time Frame: At 1 month Post intervention (survey was sent at 30 days after the last couching session)
Population: Change in the question regarding activity (t-test) between the pre and the post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 12
scores on a scale | -0.33 (0.89)

8. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Nutrition
Description: Quality of life concerning nutrition (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the 1-month post intervention survey
Time Frame: At 1 month Post intervention (survey was sent at 30 days after the last couching session)
Population: Change in the question regarding activity (t-test) between the pre and the post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 12
scores on a scale
  5-10 servings of fruits/day | 0.45 (1.51)
  Avoiding fast food | 0.36 (1.96)

9. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Sleep
Description: Quality of life concerning sleep (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre-intervention survey and 3-month post intervention survey
Time Frame: At 3 month Post intervention (survey was sent at 90 days after the last couching session)
Population: Change in the question regarding sleep (t-test) between the pre and the 3-month post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 10
scores on a scale
  7-8 hours of sleep/day: number analyzed (Participants) | 8
  7-8 hours of sleep/day | -0.63 (1.51)
  Waking up rested | -0.80 (1.55)

10. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Activity
Description: Quality of life concerning activity (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the 3-month post intervention survey
Time Frame: At 3 month Post intervention (survey was sent at 90 days after the last couching session)
Population: Change in the question regarding activity (t-test) between the pre and the 3-month post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 10
scores on a scale
  Remaining physically active | 0.70 (0.95)
  Needing help with everyday activities | -0.80 (1.48)

11. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Purpose
Description: Quality of life concerning feeling of purpose (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the 3-month post intervention survey
Time Frame: At 3 month Post intervention (survey was sent at 90 days after the last couching session)
Population: Change in the question regarding activity (t-test) between the pre and the 3- month post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 9
scores on a scale | -0.22 (0.44)

12. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Nutrition
Description: Quality of life concerning nutrition (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the 3-month post intervention survey
Time Frame: At 3 month Post intervention (survey was sent at 90 days after the last couching session)
Population: Change in the question regarding activity (t-test) between the pre and the 3- month post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 9
scores on a scale
  5-10 servings of fruits/day | 0.44 (1.81)
  Avoiding fast food | 0.89 (2.42)

13. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Resilience
Description: Quality of life concerning resilience (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the post intervention survey
Time Frame: Post intervention (survey completed at the end of last coaching session)
Population: Change in the question regarding sleep (t-test) between the pre and the post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 16
scores on a scale
  Adapting to changes | 0.00 (0.63)
  Bouncing back from illness/injury and hardship: number analyzed (Participants) | 15
  Bouncing back from illness/injury and hardship | -0.13 (0.64)

14. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Resilience
Description: Quality of life concerning resilience (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the 1-month post intervention survey
Time Frame: At 1 month Post intervention (survey was sent at 30 days after the last couching session)
Population: Change in the question regarding sleep (t-test) between the pre and the post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 12
scores on a scale
  Adapting to changes | 0.00 (0.95)
  Bouncing back from illness/injury and hardship: number analyzed (Participants) | 11
  Bouncing back from illness/injury and hardship | -0.36 (0.50)

15. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Resilience
Description: Quality of life concerning resilience (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the 3-month post intervention survey
Time Frame: At 3 month Post intervention (survey was sent at 90 days after the last couching session)
Population: Change in the question regarding sleep (t-test) between the pre and the 3-month post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 9
scores on a scale
  Adapting to changes | 0.00 (0.87)
  Bouncing back from illness/injury and hardship | -0.11 (0.33)

16. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Empowerment
Description: Quality of life concerning Empowerment (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the post intervention survey
Time Frame: Post intervention (survey completed at the end of last coaching session)
Population: Change in the question regarding sleep (t-test) between the pre and the post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 16
scores on a scale
  Knowledge to manage own health: number analyzed (Participants) | 15
  Knowledge to manage own health | -0.13 (0.52)
  Being in control of own health and well-being | -0.25 (1.13)
  Knowing where to turn in times of crisis/stress | -0.13 (1.09)

17. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Empowerment
Description: Quality of life concerning Empowerment (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the 1-month post intervention survey
Time Frame: At 1 month Post intervention (survey was sent at 30 days after the last couching session)
Population: Change in the question regarding sleep (t-test) between the pre and the 1-month post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 12
scores on a scale
  Knowledge to manage own health | -0.33 (0.49)
  Being in control of own health and well-being | -0.33 (0.49)
  Knowing where to turn in times of crisis/stress | -0.25 (1.14)

18. Primary Outcome: Change in Quality of Life Post Intervention (Coaching Sessions) - Empowerment
Description: Quality of life concerning Empowerment (on 1-5 Likert scale with 1 being the worst and 5 the best in each category) developed for this project.
  Change between the pre and the 3-month post intervention survey
Time Frame: At 3 month Post intervention (survey was sent at 90 days after the last couching session)
Population: Change in the question regarding sleep (t-test) between the pre and the 1-month post intervention survey
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Personal Resilience Empowerment Program
Number analyzed (Participants) | 10
scores on a scale
  Knowledge to manage own health | -0.20 (0.42)
  Being in control of own health and well-being | -0.40 (0.70)
  Knowing where to turn in times of crisis/stress: number analyzed (Participants) | 9
  Knowing where to turn in times of crisis/stress | -0.22 (0.83)

ADVERSE EVENTS:
Time Frame: 3 months post-op
Description: Any adverse events related to the Personal Resilience Empowerment Program Study
Groups:
- Personal Resilience Empowerment Program (All Visits and Follow up): Participants who were enrolled, completed all visits and completed the two follow-up visits (1 month and 3 months post-op)
- Personal Resilience Empowerment Program (Visits Only): Participants who were enrolled and completed the first three visits (but not follow-up)
Arm/Group | Personal Resilience Empowerment Program (All Visits and Follow up) | Personal Resilience Empowerment Program (Visits Only)
All-Cause Mortality (participants affected / at risk) | 0/10 | 2/16
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/16
Other Adverse Events (participants affected / at risk) | 0/10 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Personal Resilience Empowerment Program (All Visits and Follow up) (N=10) | Personal Resilience Empowerment Program (Visits Only) (N=16)
Death due to underlining cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) — Unrelated to the Personal Resilience Empowerment Program Study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT03644173/Prot_SAP_000.pdf